CLINICAL TRIAL: NCT01008735
Title: Observational Retrospective Study to Evaluate the Incidence of the Gonadal Toxicity in Women of Reproductive Age With Hodgkin Lymphoma
Brief Title: Gonadal Toxicity in Women With Hodgkin Lymphoma
Acronym: FertHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Massimo Federico, Gruppo Italiano Studio Linfomi
Other Study IDs: FertHD
Record Dates: First submitted 2009-11-03; First posted 2009-11-06 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women with hodgkin lymphoma treated with chemotherapy

SUMMARY:
The Gruppo Italiano Studio Linfomi has been collecting data on patients with Hodgkin Lymphoma (HL) since 1988. This archive represents a homogeneous series of consecutive patients with HL. The very long follow up and the availability of clinical and treatment data make it feasible to perform a study on the gonadal toxicity related to treatment for HL.

ELIGIBILITY:
Inclusion Criteria:

* Female patients in complete remission after chemotherapy for Hodgkin lymphoma
* Age ≥ 18 e < 40 years
* Previous regular menstrual cycle
* No previous or concomitant gynecological diseases affecting reproducing function
* No other chemo-radiotherapy for other neoplasm
* Written informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients with Hodgkin lymphoma diagnosed until 2007 in Italy will be considered eligible for this study. Cases will be identified from the archives of GISL.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-07

PRIMARY OUTCOMES:
incidence of gonadal toxicity in terms of irreversible amenorrhea and infertility, in women of reproductive age with Hodgkin lymphoma treated with chemotherapy. | from end of treatment until date of last contact/visit

SECONDARY OUTCOMES:
role of a prophylactic treatment with oral contraceptives and GnRH analogs in preventing gonadal damage | from end of treatment until date of last contact/visit

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Angrilli, MD, Study Chair — GISL; Simona Falorio, MD, Study Chair — GISL; Massimo Federico, MD, Study Chair — GISL
Locations (1):
- Gruppo Italiano Studio Linfomi, Modena, Italy